CLINICAL TRIAL: NCT04010864
Title: Real-world Effectiveness and Safety of Antipsychotics in Individuals at Clinical High-risk for Psychosis: Study Protocol for a Prospective Observational Study (SHARP-2)
Brief Title: A Study of Antipsychotics in Individuals at Clinical High-risk for Psychosis (the SHARP-2 Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government); National Natural Science Foundation of China (Other Government); Shanghai Municipal Science and Technology Commission (Other Government); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tianhong ZHANG, associate research fellow, Shanghai Mental Health Center
Other Study IDs: CRC2018ZD04
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Clinical High-risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SHARP-2: ShangHai At Risk for Psychosis-Phase 2
  Interventions: Other: routine clinical treatment

INTERVENTIONS:
Other: routine clinical treatment — Participants will be informed that this is not a treatment study and it involves naturalistic follow-up without any extra intervention. They will otherwise follow the routine clinical treatment procedure.

SUMMARY:
The current study will improve knowledge on the effectiveness and safety of the use of antipsychotics at the prodromal phase and on factors influencing the outcome, and will eventually facilitate optimisation of individualised interventions for psychosis prevention and treatment.

DETAILED DESCRIPTION:
Help-seeking first-visit participants will be consecutively recruited. Every participant meeting the inclusion criteria will be fully informed of the study and asked to sign the written informed consent before enrolment.

Two senior nurses that will conduct the initial screenings were employed to collect all diagnostic and medication information from medical records on every follow-up visit. The four psychiatrists are qualified and well-trained and will conduct the SIPS/SOPS interview at baseline and follow-up.

The investigators will systematically record medication information. A model will be established to correlate antipsychotics with clinical and functional outcomes and demonstrate whether antipsychotics are useful and safe for preventing CHR individuals from converting to psychosis.

Based on experience from the sampling process in the SHARP-1 project, the investigators will recruit 600 participants at CHR. Considering a dropout rate of 20%, 510 cases of CHR will be followed up. According to the sample size calculation formula in superiority clinical trials of new drugs, the sample size of 600 cases is adequate for the demonstration of the effectiveness and safety of antipsychotics in CHR subjects.

ELIGIBILITY:
Inclusion Criteria:

* be aged 14 to 45-year-old
* have had at least 6-years of primary education
* be drug-naïve
* be understanding the survey, be willing to enrol in the study and sign the informed consent
* Through the Structured Interview for Prodromal Syndromes/Scale of Prodromal Symptoms (SIPS/SOPS), the participants should meet the Criteria of Prodromal Syndrome. Participants should fulfil at least one of the prodromal syndrome criteria: (1) brief intermittent psychotic syndrome, (2) attenuated positive symptom syndrome, or (3) genetic risk and deterioration syndrome

Exclusion Criteria:

* Through the Mini-International Neuropsychiatric Interview (MINI), Axis I mental disorders such as schizophrenia, affective disorders, and anxiety spectrum disorders will be excluded
* Acute or chronic renal failure; liver cirrhosis or active liver diseases
* Abnormal laboratory tests results judged by the researchers to be clinically significant and considered to affect the efficacy of the test drugs or the safety of the subjects
* Severe or unstable physical diseases, including: neurological disorders (delirium, dementia, stroke, epilepsy, migraine, etc.), congestive heart failure, angina pectoris, myocardial infarction, arrhythmia, hypertension (including untreated or uncontrolled hypertension), malignant tumours, immune compromise, and blood glucose above 12 mmol/L
* Alcohol abuse within 30 days, or alcohol or drug dependence within 6 months before the trial
* Pregnant or lactating women, or women in childbearing age who are positive in urine human chorionic gonadotropin test, or men and women who do not take effective contraceptive measures or plan for pregnancy within 3 months after the initiation of the trial
* Stroke within the last month
* Participating in any clinical trial within 30 days before the baseline
* Other situations judged by the investigators not to be suitable for the clinical trial

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Help-seeking first-visit participants will be consecutively recruited from the Shanghai Psychotherapy and Psychological Counselling Centre at the Shanghai Mental Health Centre. They will be screened for eligibility by their clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Conversion to psychosis | 4 weeks
  It will be determined using the criteria for the Presence of Psychotic Symptoms from SIPS. Specifically, the conversion will be defined by the presence of level 6 positive symptoms (the rating "6" refers to severe and psychotic symptoms) identified as either dangerous, disorganised, or occurring at least one hour a day on average, over four days a week for at least 16 hours.
Poor function | 4 weeks
  It will be determined by GAF score. Specifically, poor function outcome is defined as the GAF score of less than 60 at the follow-up point.

CONTACTS AND LOCATIONS:
Overall Officials: TianHong Zhang, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Fusar-Poli P, Borgwardt S, Bechdolf A, Addington J, Riecher-Rossler A, Schultze-Lutter F, Keshavan M, Wood S, Ruhrmann S, Seidman LJ, Valmaggia L, Cannon T, Velthorst E, De Haan L, Cornblatt B, Bonoldi I, Birchwood M, McGlashan T, Carpenter W, McGorry P, Klosterkotter J, McGuire P, Yung A. The psychosis high-risk state: a comprehensive state-of-the-art review. JAMA Psychiatry. 2013 Jan;70(1):107-20. doi: 10.1001/jamapsychiatry.2013.269. PMID 23165428
- [Background] Nelson B, Yuen HP, Wood SJ, Lin A, Spiliotacopoulos D, Bruxner A, Broussard C, Simmons M, Foley DL, Brewer WJ, Francey SM, Amminger GP, Thompson A, McGorry PD, Yung AR. Long-term follow-up of a group at ultra high risk ("prodromal") for psychosis: the PACE 400 study. JAMA Psychiatry. 2013 Aug;70(8):793-802. doi: 10.1001/jamapsychiatry.2013.1270. PMID 23739772
- [Background] Lindstrom E, Bingefors K. Patient compliance with drug therapy in schizophrenia. Economic and clinical issues. Pharmacoeconomics. 2000 Aug;18(2):106-24. doi: 10.2165/00019053-200018020-00002. PMID 11067646
- [Background] Crumlish N, Whitty P, Clarke M, Browne S, Kamali M, Gervin M, McTigue O, Kinsella A, Waddington JL, Larkin C, O'Callaghan E. Beyond the critical period: longitudinal study of 8-year outcome in first-episode non-affective psychosis. Br J Psychiatry. 2009 Jan;194(1):18-24. doi: 10.1192/bjp.bp.107.048942. PMID 19118320
- [Background] Zhang T, Xu L, Tang Y, Cui H, Wei Y, Wang J, Tang X, Li C, Wang J. Duration of untreated prodromal symptoms in a Chinese sample at a high risk for psychosis: demographic, clinical, and outcome. Psychol Med. 2018 Jun;48(8):1274-1281. doi: 10.1017/S0033291717002707. Epub 2017 Nov 27. PMID 29173206
- [Background] Zhang T, Xu L, Tang Y, Cui H, Tang X, Wei Y, Wang Y, Hu Q, Qian Z, Liu X, Li C, Wang J. Relationship between duration of untreated prodromal symptoms and symptomatic and functional recovery. Eur Arch Psychiatry Clin Neurosci. 2019 Dec;269(8):871-877. doi: 10.1007/s00406-018-0917-z. Epub 2018 Jun 25. PMID 29942980
- [Background] Zhang T, Cui H, Wei Y, Tang Y, Xu L, Tang X, Zhu Y, Jiang L, Zhang B, Qian Z, Chow A, Liu X, Li C, Xiao Z, Wang J. Progressive decline of cognition during the conversion from prodrome to psychosis with a characteristic pattern of the theory of mind compensated by neurocognition. Schizophr Res. 2018 May;195:554-559. doi: 10.1016/j.schres.2017.08.020. Epub 2017 Aug 18. PMID 28823722
- [Background] Zhang T, Cui H, Tang Y, Xu L, Li H, Wei Y, Liu X, Chow A, Li C, Jiang K, Xiao Z, Wang J. Correlation of social cognition and neurocognition on psychotic outcome: a naturalistic follow-up study of subjects with attenuated psychosis syndrome. Sci Rep. 2016 Oct 10;6:35017. doi: 10.1038/srep35017. PMID 27721394
- [Background] Collin G, Seidman LJ, Keshavan MS, Stone WS, Qi Z, Zhang T, Tang Y, Li H, Anteraper SA, Niznikiewicz MA, McCarley RW, Shenton ME, Wang J, Whitfield-Gabrieli S. Functional connectome organization predicts conversion to psychosis in clinical high-risk youth from the SHARP program. Mol Psychiatry. 2020 Oct;25(10):2431-2440. doi: 10.1038/s41380-018-0288-x. Epub 2018 Nov 8. PMID 30410064
- [Background] Shakory S, Watts JJ, Hafizi S, Da Silva T, Khan S, Kiang M, Bagby RM, Chavez S, Mizrahi R. Hippocampal glutamate metabolites and glial activation in clinical high risk and first episode psychosis. Neuropsychopharmacology. 2018 Oct;43(11):2249-2255. doi: 10.1038/s41386-018-0163-0. Epub 2018 Jul 28. PMID 30087434
- [Background] Rauchensteiner S, Kawohl W, Ozgurdal S, Littmann E, Gudlowski Y, Witthaus H, Heinz A, Juckel G. Test-performance after cognitive training in persons at risk mental state of schizophrenia and patients with schizophrenia. Psychiatry Res. 2011 Feb 28;185(3):334-9. doi: 10.1016/j.psychres.2009.09.003. Epub 2010 May 21. PMID 20493540
- [Background] Amminger GP, Schafer MR, Papageorgiou K, Klier CM, Cotton SM, Harrigan SM, Mackinnon A, McGorry PD, Berger GE. Long-chain omega-3 fatty acids for indicated prevention of psychotic disorders: a randomized, placebo-controlled trial. Arch Gen Psychiatry. 2010 Feb;67(2):146-54. doi: 10.1001/archgenpsychiatry.2009.192. PMID 20124114
- [Background] McGorry PD, Nelson B, Markulev C, Yuen HP, Schafer MR, Mossaheb N, Schlogelhofer M, Smesny S, Hickie IB, Berger GE, Chen EY, de Haan L, Nieman DH, Nordentoft M, Riecher-Rossler A, Verma S, Thompson A, Yung AR, Amminger GP. Effect of omega-3 Polyunsaturated Fatty Acids in Young People at Ultrahigh Risk for Psychotic Disorders: The NEURAPRO Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):19-27. doi: 10.1001/jamapsychiatry.2016.2902. PMID 27893018
- [Background] McGorry PD, Yung AR, Phillips LJ, Yuen HP, Francey S, Cosgrave EM, Germano D, Bravin J, McDonald T, Blair A, Adlard S, Jackson H. Randomized controlled trial of interventions designed to reduce the risk of progression to first-episode psychosis in a clinical sample with subthreshold symptoms. Arch Gen Psychiatry. 2002 Oct;59(10):921-8. doi: 10.1001/archpsyc.59.10.921. PMID 12365879
- [Derived] Zeng J, Raballo A, Gan R, Wu G, Wei Y, Xu L, Tang X, Hu Y, Tang Y, Chen T, Li C, Wang J, Zhang T. Antipsychotic Exposure in Clinical High Risk of Psychosis: Empirical Insights From a Large Cohort Study. J Clin Psychiatry. 2022 Mar 21;83(3):21m14092. doi: 10.4088/JCP.21m14092. PMID 35324095